CLINICAL TRIAL: NCT06215079
Title: Investigation of the Efficacy of Transcranial Magnetic Stimulation in Patients Developing Complex Regional Pain Syndrome Type 1 in the Upper Extremity During the Subacute-Chronic Period After Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Özlem Yücealp, Research Assistant in Physical Medicine and Rehabilitation, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10028974
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Complex Regional Pain Syndromes
Keywords: complex regional pain syndrome; transcranial magnetic stimulation; ischemic stroke
MeSH Terms: conditions — Complex Regional Pain Syndromes; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active transcranial magnetic stimulation in stroke patients with complex regional pain syndrome (Active Comparator): The intermittent theta-burst stimulation (iTBS) intensity for patients, applied under doctor supervision for a total of 5 days over one week (from Monday to Friday), will be set at 70% of the resting motor threshold. Stimulation will consist of bursts at a frequency of 50 Hz, with 3 bursts every 10 seconds, each burst lasting 2 seconds, totaling 600 bursts. Subsequently, the resting motor threshold will be adjusted to 80%, and a total of 2000 bursts will be delivered at a frequency of 10 Hz, repeated every 30 seconds, each lasting 10 seconds.
  Interventions: Device: The Magstim Rapid2 Plus Magnetic Stimulator (Magstim, Whitland, Dyfed, UK)
- sham transcranial magnetic stimulation in stroke patients with complex regional pain syndrome (Sham Comparator): Similar protocol will be applied and sham transcranial magnetic stimulation treatment will be given with a sham coil to the sham group.
  Interventions: Device: Sham transcranial magnetic stimulation
- conventional rehabilitation program in stroke patients with complex regional pain syndrome (Placebo Comparator): Only a conventional rehabilitation program consisting of discontinuous ultrasound, transcutaneous electrical nerve stimulation (TENS), and contrast bath, formed by 5 sessions, will be applied to this group.
  Interventions: Device: conventional rehabilitation program

INTERVENTIONS:
Device: The Magstim Rapid2 Plus Magnetic Stimulator (Magstim, Whitland, Dyfed, UK) — Transcranial Magnetic Stimulation (rTMS) is a non-invasive brain stimulation method that modulates the cortical excitability of the targeted motor area. While single-pulse TMS is generally used to explore the functioning of the brain, repetitive TMS is employed to induce lasting changes in brain activity. High-frequency rTMS leads to an increase in excitability in the motor cortex, whereas low-frequency application results in inhibition of motor cortical excitability. Theta-burst stimulation (TBS) is a form of rTMS that can be delivered continuously (cTBS) or intermittently (iTBS), thus modulating the excitability of corticospinal neurons beneath the stimulation area to either decrease or increase. rTMS is a growing research area in pain management, proven to be a safe and well-tolerated method. Studies have shown that rTMS applied to the motor cortex is a promising treatment method for chronic pain
  Arms: active transcranial magnetic stimulation in stroke patients with complex regional pain syndrome
Device: Sham transcranial magnetic stimulation — Patients in the control group will receive sham transcranial magnetic stimulation with sham coil for 35 minutes a day, 5 sessions in total, together with conventional rehabilitation.
  Arms: sham transcranial magnetic stimulation in stroke patients with complex regional pain syndrome
Device: conventional rehabilitation program — Patients will receive 5 minutes of continuous ultrasound (1MHz, 2W/cm2, 1:4)), followed by a 20-minute contrast bath, and 15 minutes of TENS (frequency: 100 Hz; pulse duration: 50-100 ms; and amplitude adjusted to avoid discomfort or muscle contraction to the patient).
  Arms: conventional rehabilitation program in stroke patients with complex regional pain syndrome

SUMMARY:
The aim of our study is to investigate transcranial magnetic stimulation (TMS) as a treatment option in Complex Regional Pain Syndrome, disseminate it to a broader patient population, and simultaneously demonstrate its applicability in the treatment of complex regional pain syndrome using a novel frequency matching.

DETAILED DESCRIPTION:
After ischemic stroke in the subacute to chronic period, 45 patients developing complex regional pain syndrome in the upper extremity will be divided into three groups: those receiving combined rTMS with conventional rehabilitation (occupational therapy and transcutaneous electrical stimulation for pain), those receiving sham rTMS with conventional rehabilitation, and those undergoing only conventional rehabilitation. The TMS group is planned to include 15 patients, the sham group 15 patients, and the group included in the conventional rehabilitation program only will also consist of 15 patients.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Complex Regional Pain Syndrome Diagnosis of ischemic stroke

Exclusion Criteria:

Epilepsy Pregnancy Cardiac Pacemaker, Brain pacemaker, Cochlear Implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Before the treatment, At the end of the treatment (1 week), Four weeks after the treatment
  A 10 cm Visual Analog Scale (VAS) has been used to objectively assess widespread body pain in patients. Participants use this scale to determine the intensity of their pain. While 0 represents no pain, 10 indicates the most severe pain experienced by the individual.
Brunnstrom's Hemiplegia Recovery Staging | Before the treatment, At the end of the treatment (1 week), Four weeks after the treatment
  According to Brunnstrom, the stages of recovery in patients developing paralysis due to stroke progress as follows: Stage 1, where muscles are completely flaccid; Stage 2, the emergence of muscle synergies; Stage 3, the peak of involuntary movements; Stage 4, a decrease in involuntary movements and the initiation of voluntary movements; Stage 5, the appearance of more coordinated movements; Stage 6, the disappearance of spasms and the observation of fine joint movements, approaching near-complete recovery; Stage 7, where all functions return to normal.
Stroke Specific Quality of Life Scale (SS-QoL) | Before the treatment, At the end of the treatment (1 week), Four weeks after the treatment
  The SS-QoL is an instrument specifically used to assess health-related QoL among individuals who experienced stroke. It has 49 items in 12 domains, varying from 49 to 245 points, with responses varying from 1 to 5 points. Higher values indicate better health-related QoL.

SECONDARY OUTCOMES:
Fugl Meyer Upper Extremity Assessment | Before treatment (initial), at the end, four weeks after treatment
  It assesses the upper extremity in three parts: shoulder-elbow-forearm (upper part of the arm), wrist, and hand, allowing for the evaluation of reflex activity, synergy patterns, and voluntary movement. The maximum score for the upper part of the arm is 36 points. Wrist assessment is scored out of 10 points, evaluating stability at different angles, joint range of motion, and complex movements. The maximum total score for upper extremity assessment using the Fugl-Meyer Assessment Scale is 66 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital Physical Therapy and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Gaertner M, Kong JT, Scherrer KH, Foote A, Mackey S, Johnson KA. Advancing Transcranial Magnetic Stimulation Methods for Complex Regional Pain Syndrome: An Open-Label Study of Paired Theta Burst and High-Frequency Stimulation. Neuromodulation. 2018 Jun;21(4):409-416. doi: 10.1111/ner.12760. Epub 2018 Mar 4. PMID 29504190
- [Background] Chang MC, Kwak SG, Park D. The effect of rTMS in the management of pain associated with CRPS. Transl Neurosci. 2020 Sep 28;11(1):363-370. doi: 10.1515/tnsci-2020-0120. eCollection 2020. PMID 33335776
- [Background] Nardone R, Brigo F, Holler Y, Sebastianelli L, Versace V, Saltuari L, Lochner P, Trinka E. Transcranial magnetic stimulation studies in complex regional pain syndrome type I: A review. Acta Neurol Scand. 2018 Feb;137(2):158-164. doi: 10.1111/ane.12852. Epub 2017 Oct 3. PMID 28971481
- See also: https://pubmed.ncbi.nlm.nih.gov/29504190/ — https://pubmed.ncbi.nlm.nih.gov/29504190/
- See also: https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7711855/ — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7711855/